CLINICAL TRIAL: NCT07103798
Title: Does a Microprocessor-Controlled Prosthetic Knee Joint Improve Mobility and Quality of Life in K2-Level Veteran Ambulators?
Brief Title: Effect of a Microprocessor-controlled Prosthetic Knee Joint on K2 Level Ambulators
Acronym: MPK-K2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RRD2-005-24W; RX005610 (Other Grant/Funding Number: VA RRD)
Record Dates: First submitted 2025-07-15; First posted 2025-08-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Transfemoral Amputation; Limb Loss; Limb Absence
Keywords: amputation; limb loss; limb deficiency; transfemoral; above-knee; prosthesis; knee joint

STUDY DESIGN:
Intervention Model Description: Using a cross-sectional experimental design, approximately 20 Veterans who are low functioning ambulators with unilateral, transfemoral amputations will be evaluated on two separate occasions at the Jesse Brown VA Medical Center or the Edward Hines, Jr. VA Hospital, first with their conventional NMPK and then again after a two-month accommodation period with the College Park Icon MPK.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MPK (Experimental): Subjects will be fitted with the College Park ICON MPK and permitted to accommodate for 2 months prior to data collection.
  Interventions: Other: College Park ICON
- NMPK (Active Comparator): Subjects will initially be evaluated walking on their conventional NMPK as a baseline prior to being fitted with the MPK.
  Interventions: Other: Conventional NMPK

INTERVENTIONS:
Other: College Park ICON — Subjects will be fitted and trained on the College Park ICON MPK. An accommodation period of 2 months will be provided prior to evaluation with the knee joint.
  Arms: MPK
Other: Conventional NMPK — Subjects will be tested walking with their conventional, mechanical prosthetic knee prior to being fitted with the MPK.
  Arms: NMPK

SUMMARY:
Microprocessor-controlled knees (MPKs) automatically adjust resistance or damping in the joint to improve swing- and/or stance-phase control as appropriate for the prosthesis user during gait. The purpose of this proposed investigation is to determine if there are substantial physical and psychological benefits to fitting lower functioning Veteran ambulators having transfemoral amputations with an MPK compared with a nonmicroprocessor-controlled knee (NMPK). Using a repeated-measures, cross-sectional experimental design, approximately 20 Veterans with unilateral, transfemoral amputations will be evaluated on two separate occasions at the Jesse Brown VA Medical Center or the Edward Hines, Jr. VA Hospital, first with their conventional NMPK and then again after a 2-month accommodation period with the College Park Icon MPK.

DETAILED DESCRIPTION:
Limb loss is a potentially devastating event in a person's life, often resulting in profound physical, psychological, and vocational consequences. A transfemoral amputation results in greater physical and functional impairment and an increased risk of falling in patients as compared to someone with a transtibial amputation. Furthermore, balance confidence and fear of falling appears to be a persistent and pervasive problem among lower-limb prosthesis users, which adversely affects mobility and quality of life. During the past 30 years there have been several major developments in prosthetic knee mechanisms that incorporate microprocessors to improve swing-phase characteristics and provide greater stability during stance phase. Microprocessor-controlled knees (MPKs) automatically adjust resistance or damping in the joint to improve swing- and/or stance-phase control as appropriate for the user during gait.

There are numerous reported benefits of MPKs over non-microprocessor controlled knees (NMPKs), including faster self-selected walking speeds, reduced cognitive burden while walking, fewer stumbles and falls, and increased perceptions of confidence and safety while ambulating. Nonetheless, MPKs are not typically prescribed or fitted on lower functioning ambulators, which is the activity classification of most Veteran patients.

The purpose of this proposed investigation is to determine if there are substantial physical and psychological benefits to fitting lower functioning Veteran ambulators having transfemoral amputations with an MPK compared with a NMPK. The specific aims and hypotheses of this project are:

Aim 1: To determine the effects of the College Park Icon on the mobility of unilateral, transfemoral prosthesis users. The investigators hypothesize that the MPK will enable users to 1) increase their freely-selected (i.e., normal) walking speed, and 2) walk over a wider range of speeds. Furthermore, the investigators hypothesize that 3) participants will report fewer falls with the MPK.

Aim 2: To determine the effects of the College Park Icon on the psychological well-being of unilateral, transfemoral prosthesis users. The investigators hypothesize that subjects will improve their scores on patient-reported outcome assessments including the ABC, OPUS, and PLUS-M with the MPK.

Aim 3: To determine subjects' preference for the College Park Icon compared to their conventional NMPK. At the completion of the study, the investigators will ask participants which prosthetic knee type they preferred. It's hypothesized that the majority of participants will prefer using the MPK over the NMPK. Those subjects who prefer the MPK will be permitted to keep the component in their prosthesis, while those who prefer their NMPK will have their prosthesis returned to its original configuration.

Using a cross-sectional experimental design, approximately 20 Veterans who are low functioning ambulators with unilateral, transfemoral amputations will be evaluated on two separate occasions at the Jesse Brown VA Medical Center or the Edward Hines, Jr. VA Hospital, first with their conventional NMPK and then again after a two-month accommodation period with the College Park Icon MPK.

This work is directly applicable to VHA's Patient Care Mission because the results may justify the fitting of MPKs on low-level ambulators within the VA system and substantially improve the mobility of Veterans with lower limb amputations while increasing their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, transfemoral amputation (any etiology).
* Age from 45-85 years.
* Residual limb length classified as standard (i.e., medium) to long.
* Prosthesis user for at least 1 year prior to enrolling in the study.
* K2-level classification while using their NMPK.
* Good sensation on their residual limb.
* Good skin integrity upon visual inspection.
* Presents with good socket fit based upon a standard assessment by the study prosthetist.

Exclusion Criteria:

* Bilateral leg amputations.
* Individuals with a knee disarticulation.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Walking speed | To be measured before and immediately following the 2-month accommodation period of wearing the MPK.
  Walking speed will be measured as participants walk on level ground at slow, normal and fast speeds.
Falls during walking | To be determined before and during the 2-month accommodation period of wearing the MPK
  The number of falls that occur while the subject is walking will be recorded in a daily diary.
PLUS-M | To be measured before and immediately following the 2-month accommodation period of wearing the MPK.
  The Prosthetic Limb User Survey of Mobility (PLUS-M) will be used to determine the mobility of subjects before and after fitting with the MPK. Scores range from 12-60 points, and a higher score indicates greater mobility.
Prosthetic Knee Preference | To be asked immediately following the 2-month accommodation period of wearing the MPK.
  Subjects will be asked which prosthetic knee they prefer at the completion of the study. For those that indicate preference for the MPK, they will be permitted to keep it in their prosthesis. For those that prefer the NMPK, their prosthesis will be restored to the configuration prior to beginning the study.

SECONDARY OUTCOMES:
ABC Scale | To be administered before and immediately following the 2-month accommodation period of wearing the MPK.
  The Activities-specific Balance Confidence (ABC) Scale measures the subject's confidence in not losing their balance or becoming unsteady while performing different activities. Scores range from 0-100%, where zero represents no confidence and 100 represents complete confidence in performing an activity without losing balance or becoming unsteady.
OPUS | To be administered before and immediately following the 2-month accommodation period of wearing the MPK.
  The Orthotics and Prosthetics User's Survey (OPUS) is a self-report questionnaire that can be used for quality assessment, to maintain awareness of improvement in activities, to evaluate changes in patient's functional status and quality of life, and to assess satisfaction with devices and services. Scores range from 0-80 points, with a higher score indicating greater functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Gard, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: No
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. Results from this study will be freely disseminated via presentations at professional conferences and publications in scientific journals. Additionally, data acquired for this project will be shared with those investigators who make a formal request to the PI and can demonstrate a legitimate and justifiable cause for utilization of such data. All requests for these data will be discussed with the VA scientific program manager.